CLINICAL TRIAL: NCT01587209
Title: Phase 1 Study Investigating Alterations of Circulating Microparticles in Scuba Divers With Decompression Sickness
Brief Title: Microparticles in Scuba Divers With Decompression Sickness
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Office of Naval Research (ONR) (U.S. Federal Agency); University of Maryland (Other)
Responsible Party: Sponsor
Other Study IDs: 814139
Record Dates: First submitted 2012-04-23; First posted 2012-04-30 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-08

CONDITIONS: Decompression Sickness; Dysbarism
Keywords: decompression; intravascular bubbles; neutrophil activation
MeSH Terms: conditions — Decompression Sickness; Barotrauma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Divers with decompression sickness: The sole group under study is SCUBA divers who have sustained decompression sickness

SUMMARY:
The investigators hypothesize that membrane microparticles (MPs) are liberated into the blood stream in response to decompression stress and that certain MPs characteristics initiate inflammatory responses that contribute to the clinical syndrome the investigators call decompression sickness. The research goal is to evaluate the number, type and time-course for elevations in MPs in sport SCUBA divers who present for treatment of decompression sickness. Blood samples are to be taken from consenting patients before and after they undergo treatment for decompression sickness and at a follow-up clinic visit from 1 to 3 weeks later (three samples total).

DETAILED DESCRIPTION:
Microparticles (MPs) are small membrane bound vesicles shed from the surface of a variety of cells by what appear to be well regulated processes. They are elevated in many physiological and disease states and in some instances have been associated with organ injury. Shear stress - as can be caused by intravascular bubbles - is one of the stimuli known to cause cells to release microparticles. Most sport SCUBA dives have been shown to generate intravascular bubbles - even safe dives well within limits established by the US Navy and sports authorities. The investigators have reported elevations in several sub-types of MPs in a group of individuals undergoing a well monitored series of open-water SCUBA dives. There is no information of the occurrence of MPs in injured divers. The investigators have published results using a murine model which demonstrated that mice subjected to varying decompression stresses exhibit progressive elevations in circulating MPs derived from leukocytes, erythrocytes, platelets and endothelial cells. Using novel interventions the investigators demonstrated that MPs cause intravascular neutrophil activation and inflammatory perivascular injuries. Therefore, there is pathophysiological information to suggest that one or more element of MPs (number and/or pro-inflammatory subtype) may be proximal elements that precipitate the clinical syndrome the investigators call decompression sickness.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are given the diagnosis of decompression sickness will be offered entry into this study

Exclusion Criteria:

* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: SCUBA divers over age 21 that present for evaluation of suspected decompression sickness
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2011-08; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Microparticle elevations in injured divers | four years
  We will quantify microparticles in plasma by standard flow cytometry techniques.

SECONDARY OUTCOMES:
Microparticle sub-types in injured divers | four years
  We will evaluate sub-types of microparticles to determine their cells of origin.
Neutrophil activation in injured divers | four years
  We will evaluate presence of neutrophil activation in injured divers.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen R Thom, MD,PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Thom SR, Yang M, Bhopale VM, Huang S, Milovanova TN. Microparticles initiate decompression-induced neutrophil activation and subsequent vascular injuries. J Appl Physiol (1985). 2011 Feb;110(2):340-51. doi: 10.1152/japplphysiol.00811.2010. Epub 2010 Oct 21. PMID 20966192
- [Background] Yang M, Milovanova TN, Bogush M, Uzun G, Bhopale VM, Thom SR. Microparticle enlargement and altered surface proteins after air decompression are associated with inflammatory vascular injuries. J Appl Physiol (1985). 2012 Jan;112(1):204-11. doi: 10.1152/japplphysiol.00953.2011. Epub 2011 Sep 29. PMID 21960660
- [Background] Thom SR, Milovanova TN, Bogush M, Bhopale VM, Yang M, Bushmann K, Pollock NW, Ljubkovic M, Denoble P, Dujic Z. Microparticle production, neutrophil activation, and intravascular bubbles following open-water SCUBA diving. J Appl Physiol (1985). 2012 Apr;112(8):1268-78. doi: 10.1152/japplphysiol.01305.2011. Epub 2012 Feb 9. PMID 22323646